CLINICAL TRIAL: NCT02224833
Title: Pharmacist-led Intervention to Reduce Potentially Inappropriate Prescription in Elderly and Polypharmacy Patients at Primary Care Setting (PHARM-PC) Cluster Randomized Trial
Brief Title: Inappropriate Prescription in Elderly and Polypharmacy Patients in Primary Care (PHARM-PC) Trial
Acronym: PHARM-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Comarcal de Inca (Other)
Responsible Party: Principal Investigator, Jesus Martinez Sotelo, Pharm D, Hospital Comarcal de Inca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHARM-PC
Record Dates: First submitted 2014-08-19; First posted 2014-08-25 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Elderly (People Aged 65 or More); Polypharmacy (People Under Treatment With 5 or More Drugs)
Keywords: appropriateness; elderly; polypharmacy; primary care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Pharmacist intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Pharmacist intervention — Systematic review of treatments:
  Identification of reasons for PPI.
  * Determination of recommended pharmacotherapeutic alternatives.
  * Issue recommendations for therapeutic appropriateness to the doctor (via registration on the EHR and verbal communication if deemed appropriate); that will be of 4 types: Add medicine, discontinue medicine, adjust dosage, replace medicine.
  After the medical visit (the next day) New treatment review for: Checking acceptance or rejection of the recommendations issued, review potential new prescriptions made without pharmacist recommending, and whether these new drugs lead to PIP.
  Arms: Intervention

SUMMARY:
PHARM-PC study is based on identify potentially inappropriate prescriptions (PIP) and delivery therapeutic appropriateness recommendations from the pharmacist to the physician and about drugs prescribed for elderly and polypharmacy patients in primary care. Assessment of the impact of pharmacist intervention on the appropriateness of prescribing and both health outcomes and economic outcomes will be done.

DETAILED DESCRIPTION:
Main objective:

To assess the effect of Pharmaceutical Intervention (PI) on PIP in elderly patients with polypharmacy in PC.

Secondary objectives:

2. a. Assess baseline characteristics of elderly polypharmacy patients in PC; and assess association with the possible presence of PIP.

2. b. Describe the main types and the reasons for PIP. 3. Assess impact of PI on health outcomes (morbidity and mortality). 4. Estimate the effect of IF on the cost of both drugs and healthcare resources.

Design and methods:

Prospective, multicenter, open-label, controlled and randomized by groups (clusters) clinical trail; in order to prevent contamination between Intervention Group (IG) and Control Group (CG) patients seen by the same physician.

Clusters (unit of randomization) are primary care physicians who work in public primary care health centers in Tramuntana Sector (under Hospital Comarcal de Inca). Different cluster were randomly assigned to Intervention Group (IG) or control group (CG) in the ratio 1: 1.

The study compared the effectiveness of a strategy for health care to elderly patients with polypharmacy in PC consisting of medical visit along with PI, consistent in turn on identifying PIP and delivering therapeutic appropriateness recommendations against routine health care, consisting solely of medical visit.

Furthermore the impact of treatment on health outcomes, and both drug and health service costs will also be assessed.

Methodology:

Intervention Group:

* Systematic review of treatments:

  * Identification of reasons for PPI: Causes why a pharmacological prescription (drug, dose, route of administration, duration of treatment) may have both risk-benefit balance as cost-effectiveness balance unfavorable versus other alternatives, such as:
* contraindications, dosage (dose, frequency, duration, inappropriate), duplication, interactions, risk of adverse effects, health problem insufficiently treated, unnecessary medication; equivalent to Drug-Related Problems (DRP) listed in the Third Consensus of Granada. To identify DRP we will use a combination of explicit criteria (STOPP / START) and implicit criteria (information from: drug labels, drug-surveillance alerts issued by drug regulatory agencies, recommendations of scientific societies); implemented in CheckTheMeds® software.
* Drugs that have more cost-effective alternatives, ranked by the Committee on Quality Indicators Prescription Health Service of the Balearic Islands as:

  * New drugs with little or no therapeutic value: drugs marketed in the past 5 years and considered by the "Comité Mixto de Evaluación de Nuevos Medicamentos" as little or no therapeutic value against the alternatives available in the market for the treatment of these pathologies: metformin / saxagliptin, linagliptin / metformin, saxagliptin, linagliptin, rosuvastatin, pitavastatin, sinecatequin, ingenol mebutate, bazedoxifene, silodosin, degarelix, denosumab, hydromorphone, tapentadol, agomelatine, desvenlafaxine, indacaterol, ciclesonide, aclidinium bromide, glycopyrronium bromide, roflumilast, bilastine, tafluprost.
  * Medications considered first choice in the treatment of the most prevalent diseases in the outpatient setting: Omeprazole (antiulcer); Metformin (oral antidiabetic); ACE inhibitors; Beta-blockers; diuretics; Calcium-antagonists (anti-hypertensive); Simvastatin (statins); diclofenac; Diclofenac / Misoprostol; ibuprofen; Naproxen (anti-inflammatory drugs); Alendronic acid (osteoporosis); fluoxetine; citalopram; paroxetine; Sertraline (antidepressant).
* Determination of recommended pharmacotherapeutic alternatives.
* Issue recommendations for therapeutic appropriateness to the doctor (via registration on the EHR and verbal communication if deemed appropriate); that will be of 4 types: Add medicine; discontinue medicine; adjust dosage; replace medicine.
* After the medical visit (the next day): New treatment review for: checking acceptance or rejection of the recommendations issued; and review potential new prescriptions made without pharmacist recommending, and whether these new drugs lead to PIP.

Control Group: In the control group, the same steps will be followed than intervention group; excluding issue recommendations for therapeutic appropriateness to the doctor.

Sample size and statistical power:

The sample size was calculated by comparing proportions using the application for the determination of sample size available on Fisterra website; based on the results of a pilot study, not yet published, which showed a difference of 15 percent in the number of patients with PIP between IG and CG and based on the study by Delgado et al, which considers cost effective any screening tool that achieves at least a moderate reduction (10-20 percent) of PIP. For a power of 80%, and assuming a loss rate of 10 percent; was obtained a sample size of 153. Considering adjustment for cluster effect, according to the following formula: 1 + (m - 1) x ρ, we obtain a final sample size of 214 patients.

Statistics:

* Categorical variables (qualitative): Measurements of frequency and percentage. The association between categorical variables will be performed by chi-square or Fischer's exact test; accordingly.
* Continuous Variables (Quantitative): Measures of central tendency and dispersion measures. The association between continuous variables will be performed using T-Student t test; ANOVA; Mann-Whitney or Kruskal-Wallis, as appropriate.

A value of p ≤ 0.05 as statistically significant will be considered.

Timescale:

The study will begin in October 2014 and will end about April 2016. Is expected than patients will be enrolled into the study between October 2014 and April 2015, until complete sample size required.

The study will last 12 more months to assess the outcomes of morbidity, mortality and cost of health care resources

Ethics and safety:

The Research Ethics Committee and Primary Care Research Unit of Balearic Islands have approved the project.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years
* treatment with 5 or more chronic medications.

Exclusion Criteria:

* routine monitoring is carried out in private health care
* temporary displaced persons (routine monitoring is carried out in another community).
* Institutionalized patients
* Patients in the Home Care Program

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 549 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with potentially inappropriate prescriptions (PIP) | Up to 6 months
  This variable will be measured six months after intervention, when a new review of patient treatment will be performed to check acceptance by the physician of the recommendations issued by the pharmacist.
  PIP: Prescription (drug, dose, frequency of administration) that meets at least one of the following conditions: contraindication, inadequate dosing (dose, frequency and / or duration), duplication, interactions, probability of adverse drug reactions, health problem insufficiently treated, unnecessary medication; new drugs of little-no therapeutic value, drug which is not considered as first choice in the treatment of the most prevalent diseases in the outpatient setting.
Mean number of PIP per patient | Up to 6 months
  This variable will be measured six months after intervention, when a new review of patient treatment will be performed to check acceptance by the physician of the recommendations issued by the pharmacist.

SECONDARY OUTCOMES:
Morbidity | Up to 12 months
  Composite end-point:
  * Hospital Admissions (HA) +
  * Visits to Hospital Emergency Department (HED) +
  * Visit to Primary Care Emergency Department (PCED) +
  * Specialized Care Consultation (SCC) +
  * Primary Care Consultations (PCC).
Total spending on drugs | Up to 6 months
  Total monetary amount (in euros) of the drugs involved in the PIP; which is calculated as annual amount (being chronic medications), for which we will consider the invoice price (monetary amount paid by the health administration for drugs) specified in the pharmaceutical sales database from Balearic Islands and total daily dose prescribed.
  This variable will be measured six months after intervention (same timeline as primary outcome), when a new review of patient treatment will be performed to check acceptance by the physician of the recommendations issued by the pharmacist.
Total spending on health resources. | Up to 12 months
  Composite end-point:
  Total monetary amount (in euros) of the following health resources used due to PIP:
  * Hospital Admissions (HA) +
  * Visits to Hospital Emergency Department (HED) +
  * Visit to Primary Care Emergency Department (PCED) +
  * Specialized Care Consultation (SCC) +
  * Primary Care Consultations (PCC). according to the survey of prices paid by the Balearic Islands Health Service to healthcare facilities arranged by provision of healthcare resources; published in the Official Gazette of the Balearic Islands.
Mortality | Up to 12 months
  Number of patients who died

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Martínez, Pharm D, Principal Investigator — Hospital Comarcal de Inca
Locations (1):
- Sector Sanitario Tramuntana, Inca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simo Minana J. [Use of prescription drugs in Spain and Europe]. Aten Primaria. 2012 Jun;44(6):335-47. doi: 10.1016/j.aprim.2011.06.009. Epub 2011 Oct 22. Spanish. PMID 22018798
- [Background] Hill-Taylor B, Sketris I, Hayden J, Byrne S, O'Sullivan D, Christie R. Application of the STOPP/START criteria: a systematic review of the prevalence of potentially inappropriate prescribing in older adults, and evidence of clinical, humanistic and economic impact. J Clin Pharm Ther. 2013 Oct;38(5):360-72. doi: 10.1111/jcpt.12059. Epub 2013 Apr 2. PMID 23550814
- [Background] Gallagher P, Ryan C, Byrne S, Kennedy J, O'Mahony D. STOPP (Screening Tool of Older Person's Prescriptions) and START (Screening Tool to Alert doctors to Right Treatment). Consensus validation. Int J Clin Pharmacol Ther. 2008 Feb;46(2):72-83. doi: 10.5414/cpp46072. PMID 18218287
- See also: Tercer Consenso de Granada sobre Problemas Relacionados con Medicamentos (PRM) y Resultados Negativos asociados a la Medicación (RNM). Ars Pharm, 48(1), 5-17 — http://farmacia.ugr.es/ars/pdf/374.pdf